CLINICAL TRIAL: NCT01609660
Title: Impact of Probiotics on the Intestinal Microbiota and Its Association With Postoperative Outcome After Colorectal Surgery
Brief Title: Impact of Probiotics on the Intestinal Microbiota
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Maria Isabel Toulson Davisson Correia, Professor of Surgery, responsible investigator, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDS - APQ-01005-11; CDS - APQ-01005-11 (Other Grant/Funding Number: FAPEMIG - CDS - APQ-01005-11)
Record Dates: First submitted 2012-05-27; First posted 2012-06-01 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Cancer
Keywords: probiotics; cytokine; short chain fatty acids; complications; colorectal surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): No intervention at all
- Study group (Experimental): Use of Saccharomyces boulardii, 100mg for at least seven days before surgery
  Interventions: Dietary Supplement: Saccharomyces boulardii

INTERVENTIONS:
Dietary Supplement: Saccharomyces boulardii — 100mg daily for seven days prior to surgery
  Other Names: Floratil
  Arms: Study group

SUMMARY:
The purpose of this study is to assess the impact of probiotic administration (Saccharomyces boulardii) on patients undergoing colorectal resections comparing to the routine protocol by assessing: (1)intestinal microbiota modulation using RT-PCR to measure cytokine in the mucosa; (2) assess postoperative complications, mainly infectious and mortality, as well as length of hospital stay

DETAILED DESCRIPTION:
The intestinal microbiota, a complex and dynamic population of different bacterial species, under normal circumstances, represents an important contribution to the health of the host. This plays a key role by maintaining the integrity of the epithelial barrier and helping the development of mucosal immunity. However, under some stressful situations, such as after gastrointestinal surgery, infectious complications may be originated from the patient's own intestinal microbiota. This leads to the so called "gut origin of sepsis" hypothesis. On the other hand, under similar conditions, the supply of probiotics, the good bacteria, has been shown to be beneficial, despite few controversial results. Therefore, it is important to carefully assess the efficacy of probiotics in the prevention and treatment of complications in surgical patients, as well as to evaluate the safety of its use.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old
* intend to undergo elective colon resection at the UFMG Hospital

Exclusion Criteria:

* Patients in use of steroids
* Patients unable to receive the probiotics for, at least, 7 days before the operation
* Changes to the operation strategy
* Patients that discontinued probiotic use
* Patients who had previously taken any probiotic or prebiotic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Mucosal cytokine | April 2013
  To assess mucosal cytokine levels

SECONDARY OUTCOMES:
Short chain fatty acids | April 2013
  Assess mucosal short chain fatty acids

CONTACTS AND LOCATIONS:
Overall Officials: Maria Isabel Correia, MD, PhD, Principal Investigator — UFMG

IPD SHARING:
Plan to Share IPD: Yes
Scientific publications